CLINICAL TRIAL: NCT04233138
Title: Optimizing Therapies and Technologies to Reduce Hypoglycemia in Type 1 Diabetes Through the SUPPORT Online Platform for Self-management Education and Support
Brief Title: SUPPORT Online Training Platform for Type 1 Diabetes Self-management Education and Support (SUPPORT)
Acronym: SUPPORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Institut de Recherches Cliniques de Montreal (Other); Juvenile Diabetes Research Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Anne-Sophie Brazeau, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SUPPORT
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2022-04

CONDITIONS: Type 1 Diabetes Mellitus With Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Participants enrolling in the study have access to the online platform for 12 months (6 months with reminders, 6 months no reminders).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): The intervention group will have immediate access to the SUPPORT platform.
  Interventions: Other: SUPPORT online platform for people with type 1 diabetes

INTERVENTIONS:
Other: SUPPORT online platform for people with type 1 diabetes — All participants accepting the SUPPORT study will receive the full intervention for 6 months. Their learning is individualized depending on the way they take their insulin (injection or pump) and the way they measure their blood sugar (finger prick or continuous glucose monitoring).
  The training program starts with mandatory module on hypoglycemia. Once completed, participants will unlock all level 1 (out of 3 levels) modules from the 6 categories (medication, blood sugar monitoring, nutrition, physical activity, hypo- and hyperglycemia, health and other situations). The platform contains functionalities such as discussion forum, quizzes, videos, downloadable forms, etc. During the first 6 months, participants will receive a bi-weekly newsletter to inform them about what's new on the platform.

SUMMARY:
There are evidences that some healthcare teams are not proposing new therapeutic and technology options that have the potential to reduce hypoglycemia for people with type 1 diabetes. In practice, people living with type 1 diabetes report receiving education related to insulin pumps usage mainly on key functions (how the device works) at initiation and not enough about proactive adjustments (how to optimally use the device) especially on the long-term. In brief, short-term education is technical and product-specific, rather than being based on patients' needs.There is a need to test the efficacy of different programs that may be more suited to patients' needs and desires while offering the opportunity to reduce costs (e.g. web based). Since there is a lack of expertise related to optimal use of new technologies and therapies for people living with type 1 diabetes, we propose to design and test a web-based training (e.g. courses including videos and quizzes) and support (e.g. discussion forum) platform. This will be tested through a registry-based trial.

The overall purpose of this study is to evaluate, among a group of adults living with type 1 diabetes, the SUPPORT online education platform in terms of users' satisfaction, engagement and efficacy to change the fear and the frequency of hypoglycemia.

DETAILED DESCRIPTION:
Design and development of the SUPPORT platform:

The SUPPORT platform was designed based on the Behavior change wheel framework. The research team identified the main barriers in achieving adequate blood glucose management and in the use of an online training platform; then, features (downloadable PDFs, videos, quizzes, etc.) were designed to overcome these barriers. These training modules were developed by a team including two dietitians/certified diabetes educator, a nurse, a psychologist and endocrinologist (all specialized in type 1 diabetes). The content was then reviewed by the committee of patient-partners and clinicians working in type 1 diabetes (one endocrinologist, two residents in endocrinology, two dietitians (1 being a certified diabetes educator) and two nurses (1 being a certified diabetes educator).

Recruitment and intervention:

Recruitment of people with type 1 diabetes will be done via an email sent to the participants who completed phase 2 of the BETTER registry, are 18 years old or older, and agreed to be contacted for other studies. All participants accepting to participate will receive the full intervention for 6 months (access to the platform with bi-weekly newsletters). During the following 6 months, participants will still have access to the platform, but no newsletter will be sent (sustainability phase). Questionnaires will be given at baseline, 6-month, and 12-month of the intervention to assess fear of hypoglycemia, diabetes knowledge, overall satisfaction of the platform. Participant will also receive 1 question every 6 weeks regarding the frequency of hypoglycemia during the last 3 days. The observational control group will not have access to the platform. We will extract data from the baseline, 6 months and annual registry completion.

Analysis:

Initial analysis will be descriptive and baseline data will be summarized separately for both groups. Baseline continuous data will be reported as means with standard deviations (median and interquartile range if data are skewed). Categorical data will be reported as proportions. Our primary outcome is the difference in mean self-reported hypoglycemia and fear of hypoglycemia score between the 2 groups after 6 months of intervention. The primary outcome will be calculated and compared between the two groups using differences with 95% CI using paired t-test and McNemar test. Analysis will be by intention to treat.

Sample size and pairing:

Every participant in the intervention group will be randomly paired by gender and date of completion of the phase 2 BETTER questionnaire (+/- 1 month) with a participant who answered the second phase of the BETTER registry but who did not respond to the invitation e-mail for the SUPPORT study. We have calculated the number of pairs to be able to detect a 25% reduction in adults given the small but present difference in self-reported hypoglycemia in both age groups. We estimate a 25% reduction in hypoglycemic episodes for a between-group difference of 0.95. Assuming a common standard deviation of 4.5, for a 2-sided alpha=0.05 and 80% power to detect such a difference with sample size calculation for comparing paired differences, we will require 179 pairs of participants in total. Allowing for a up to 35% loss to follow-up, we will require 275 pairs of participants.

Importance of this study:

Once validated, the SUPPORT online training platform for individuals with type 1 diabetes can be a low-cost and easily accessible training to complement regular care and increase knowledge of diabetes-related therapies and technologies.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. Completed phase 2 of the BETTER registry
3. Self-reported diagnosis of type 1 diabetes for ≥ 1 year
4. Daily use of ≥ 4 injections of insulin or CSII
5. Have access to Internet
6. Use of an active email address
7. Comprehension of English or French

Exclusion Criteria:

1. Ongoing pregnancy
2. Other illnesses limiting diabetes care or access to the platform (e.g. dementia and blindness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Users' satisfaction of the SUPPORT platform | after 6 months
  Online questionnaire- General satisfaction of the SUPPORT platform-8 items

SECONDARY OUTCOMES:
Users' engagement on the SUPPORT platform | baseline to 6 months
  Extracted from Google Analytics: Number of page viewed, time spent on the platform, number of downloaded PDFs, number of forum posts
Change in the frequency and the fear of hypoglycemia | 6-month, and 12-month
  Self-reported (compared to baseline)
Change in the glycated hemoglobin | at 6 months and 12 months
  Self-reported (compared to baseline)
Knowledge about diabetes self-management | at baseline, 6 months and 12 months
  Online questionnaire based on content seen on the SUPPORT platform- 7 items

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Brazeau, PhD, Principal Investigator — McGill University
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Xie LF, Housni A, Roy-Fleming A, Bandini A, Delormier T, Costa DD, Brazeau AS. Evaluation of Support, a self-guided online type 1 diabetes self-management education and support web application-a mixed methods study. Digit Health. 2023 Sep 28;9:20552076231204435. doi: 10.1177/20552076231204435. eCollection 2023 Jan-Dec. PMID 37780064